CLINICAL TRIAL: NCT06044207
Title: Biomarkers and Risk Factors for Perioperative Neurocognitive Disorders in Elderly Non-neurosurgical Patients
Brief Title: Biomarkers and Risk Factors for Perioperative Neurocognitive Dysfunction in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinan Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-076-01
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Neurocognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with perioperative neurocognitive dysfunction
  Interventions: Diagnostic Test: Pittsburgh sleep quality index; Diagnostic Test: Self-rating depression scale; Diagnostic Test: Montreal Cognitive Assessment
- Patients without perioperative neurocognitive dysfunction
  Interventions: Diagnostic Test: Pittsburgh sleep quality index; Diagnostic Test: Self-rating depression scale; Diagnostic Test: Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Pittsburgh sleep quality index — The scale is suitable for evaluating sleep quality in patients with sleep disorders and psychiatric disorders, as well as for assessing sleep quality in the general population.
Diagnostic Test: Self-rating depression scale — The scale is easy to use, can fairly intuitively reflect whether the patient has depression and the degree of depression, has been widely used in outpatient gross screening, mood state assessment.
Diagnostic Test: Montreal Cognitive Assessment — The scale is a tool used for rapid screening of mild cognitive dysfunction to identify patients with preoperative cognitive dysfunction

SUMMARY:
Basic information and biological samples of patients were collected preoperatively and intraoperatively, and patients were divided into case and control groups by cognitive function assessment postoperatively, and risk factors and biomarkers of perioperative cognitive dysfunction were derived by analyzing and statistically processing basic information and biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 65 years old
* ASA classification Ⅰ~Ⅲ grade

Exclusion Criteria:

* History of previous Craniocerebral surgery or Craniocerebral trauma
* Inability to successfully complete preoperative psychological function tests
* Those who are severely deaf, speech impaired and otherwise unable to communicate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people older than 65 years old who have been identified for non-neurosurgical procedures at Jinan Central Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative neurocognitive dysfunction | 1 year postoperative
  Identification of patients who develop perioperative neurocognitive disorders after surgery by postoperative follow-up with cognitive function tests

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China